CLINICAL TRIAL: NCT07191093
Title: Predictors of Right Ventricle Dysfunction After Pulmonary Balloon Valvuloplasty
Brief Title: Predictors of RV Dysfunction After BPV
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Farah Fawzy, Principal Investigator, Assiut University
Other Study IDs: RV Dysfunction post BPV
Record Dates: First submitted 2025-08-22; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-08

CONDITIONS: RV Dysfunction; Pulmonary Valvuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pulmonary valvuloplasty — Pulmonary balloon valvuloplasty (PBV) is the treatment of choice for moderate to severe valvular pulmonary stenosis. It is a minimally invasive, catheter-based intervention that involves dilation of the stenotic pulmonary valve using an appropriately sized balloon. The goal is to relieve obstruction, reduce right ventricular pressure, and prevent long-term complications such as RV hypertrophy, dysfunction, and arrhythmias. The procedure has shown excellent immediate and long-term outcomes, particularly in patients with a pliable, doming pulmonary valve and no significant regurgitation or associated congenital lesions.

SUMMARY:
This aim focuses on :

Assessing how common RV dysfunction is post-procedure Evaluating RV function changes over time (e.g., TAPSE, FAC, RV strain if available) Identifying risk factors or predictors (e.g., high residual gradient, severe PR, age at intervention)

DETAILED DESCRIPTION:
Pulmonary stenosis (PS) is a congenital or acquired narrowing of the right ventricular outflow tract (RVOT) at the level of the pulmonary valve, leading to obstruction of blood flow from the right ventricle (RV) to the pulmonary artery. It accounts for approximately 8-10% of all congenital heart diseases and occurs most commonly as an isolated valvular lesion. Valvular PS is characterized by thickened, fused, or dysplastic pulmonary valve leaflets, resulting in increased right ventricular pressure and compensatory hypertrophy. Over time, if untreated, this can progress to right ventricular dilation, dysfunction, and right-sided heart failure.

Pulmonary balloon valvuloplasty (PBV) is the treatment of choice for moderate to severe valvular pulmonary stenosis. It is a minimally invasive, catheter-based intervention that involves dilation of the stenotic pulmonary valve using an appropriately sized balloon. The goal is to relieve obstruction, reduce right ventricular pressure, and prevent long-term complications such as RV hypertrophy, dysfunction, and arrhythmias. The procedure has shown excellent immediate and long-term outcomes, particularly in patients with a pliable, doming pulmonary valve and no significant regurgitation or associated congenital lesions.

Despite the effectiveness and safety of PBV, complications can occur, and among them, right ventricular dysfunction is a critical concern. RV dysfunction post-valvuloplasty may result from several mechanisms, including longstanding pre-procedural pressure overload, myocardial fibrosis, sudden afterload reduction, procedural trauma, or development of significant pulmonary regurgitation. This dysfunction can be subtle or overt and may impact the long-term clinical outcome, exercise tolerance, and quality of life of patients.

Therefore, understanding the predictors of right ventricular dysfunction after pulmonary balloon valvuloplasty is essential. Identifying high-risk patients pre-intervention and monitoring RV function post-procedure using echocardiographic parameters such as TAPSE, fractional area change (FAC), RV strain, and tricuspid annular tissue Doppler velocity (S') can guide better management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Any age group(no age restriction) Diagnosis of isolated valvular pulmonary stenosis confirmed by echocardiographic evaluation.

Patients who have undergone or are scheduled to undergo successful pulmonary balloon valvuloplasty (PBV), defined as a post-procedural peak gradient <40 mmHg with no significant residual obstruction.

Normal or mildly dysplastic pulmonary valve morphology suitable for balloon valvuloplasty.

No history of prior cardiac surgery or transcatheter pulmonary valve intervention.

Exclusion Criteria:

* Presence of other congenital heart diseases (e.g., TOF, VSD, ASD) Previous surgical or catheter-based intervention on the pulmonary valve. Dysplastic pulmonary valve morphology not suitable for PBV Subvalvular or supravalvular pulmonary stenosis. Development of significant procedural complications, such as severe pulmonary regurgitation requiring urgent surgical intervention.

Patients in hemodynamic shock, with uncontrolled arrhythmias, or other unstable clinical conditions that may interfere with echocardiographic evaluation or follow-up.

Presence of major systemic illnesses (e.g., advanced hepatic, renal, or pulmonary disease) that could independently affect right heart function or limit follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients with isolated valvular pulmonary stenosis undergoing pulmonary balloon valvuloplasty (PBV) at the Cardiovascular Department, Assiut University Hospitals over 3 years. All ages will be included.
  Exclusion criteria: patients with subvalvular/supravalvular PS, other major congenital heart disease, previous valve intervention, hemodynamic shock, or poor echo windows.
  A minimum of 60 patients will be recruited. Clinical data, ECG, echo (including speckle tracking), and procedural details will be collected. Patients will be followed at discharge, 1 month, and 6 months to assess RV function and outcomes.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in peak transvalvular gradient after PBV | Baseline, 72 hours post-procedure, and 6 months follow-up.
Change in mean transvalvular gradient after pulmonary balloon valvuloplasty | Baseline, 72 hours post-procedure, and 6 months follow-up.
Change in estimated pulmonary artery systolic pressure PASP after PBV | Baseline, 72 hours post-procedure, and 6 months follow-up.
Change in TAPSE after PBV | Baseline, 72 hours post-procedure, and 12 months follow-up

SECONDARY OUTCOMES:
Procedural outcomes and complications | one year
  Acute procedural success (≥50% reduction in peak systolic gradient with final gradient <40 mmHg), development of pulmonary regurgitation (graded as mild, moderate, or severe), and occurrence of vascular or procedural complications (arrhythmias, balloon rupture, bleeding, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: salma mohamed taha, assistant professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Kan JS, White RI Jr, Mitchell SE, Gardner TJ. Percutaneous balloon valvuloplasty: a new method for treating congenital pulmonary-valve stenosis. N Engl J Med. 1982 Aug 26;307(9):540-2. doi: 10.1056/NEJM198208263070907. No abstract available. PMID 7099226
- [Background] Baumgartner H, De Backer J, Babu-Narayan SV, Budts W, Chessa M, Diller GP, Lung B, Kluin J, Lang IM, Meijboom F, Moons P, Mulder BJM, Oechslin E, Roos-Hesselink JW, Schwerzmann M, Sondergaard L, Zeppenfeld K; ESC Scientific Document Group. 2020 ESC Guidelines for the management of adult congenital heart disease. Eur Heart J. 2021 Feb 11;42(6):563-645. doi: 10.1093/eurheartj/ehaa554. No abstract available. PMID 32860028
- [Background] Stout KK, Daniels CJ, Aboulhosn JA, Bozkurt B, Broberg CS, Colman JM, Crumb SR, Dearani JA, Fuller S, Gurvitz M, Khairy P, Landzberg MJ, Saidi A, Valente AM, Van Hare GF. 2018 AHA/ACC Guideline for the Management of Adults With Congenital Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Apr 2;73(12):e81-e192. doi: 10.1016/j.jacc.2018.08.1029. Epub 2018 Aug 16. No abstract available. PMID 30121239
- [Background] Nasir M, Dejene K, Bedru M, Markos S. Percutaneous balloon pulmonary valvuloplasty in children: a 10-Year retrospective follow-up study in resource-limited settings. BMC Cardiovasc Disord. 2025 May 26;25(1):402. doi: 10.1186/s12872-025-04881-8. PMID 40419953